CLINICAL TRIAL: NCT01117324
Title: Bone Density of Large Newborn Infants and Infants of Diabetic Mothers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Ayala Maayan-Metzger, Sheba Medical Center
Other Study IDs: SHEBA-10-7637-AM-CTIL
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Bone Density
Keywords: Bone density; infant of diabetic mother; large birth weight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Bone density was found to be impaired among lage babies and infants of diabetic mothers as found in small group studies. The assumption is that large weight decreases fetal movements and causes decreased bone mineralization.The aim of the study is to compare 2 study groups - of large infants and infants of diabetic mothers to each other and to controls.

ELIGIBILITY:
Inclusion Criteria:

* Term infants of birth weight 4 kg and above, and
* Infants of diabetic mothers.

Exclusion Criteria:

* Preterms,
* Major congenital malformations,
* Sick babies.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Healthy term infants of birth weight 4 kg and above and infants of diabetic mothers
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Bone density | 1 week